CLINICAL TRIAL: NCT05798351
Title: Prevalence of Rectal Carriage of Carbapenemase Producing-Enterobacteriaceae on Admission to a French University Teaching Hospital
Brief Title: Rectal Carriage of Carbapenemase Producing-Enterobacteriaceae on Admission to a French University Teaching Hospital
Acronym: Prev-CPE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220938
Record Dates: First submitted 2023-01-12; First posted 2023-04-04 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Rectal Carriage of Carbapenemase Producing-Enterobacteriaceae
Keywords: Universal screening; Hospital; Rectal carriage; Enterobacteriaceae; Carbapenemase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
"The emergence and spread of highly resistant bacteria, including carbapenemase-producing Enterobacteriaceae (CPE), is a public health challenge given their rapid spread and the lack of active antibiotics against these bacteria. The spread of extended-spectrum β-lactamase-producing Enterobacteriaceae (ESBLE) since the early 2000s raises concerns about a potential similar spread of CPE in the coming years, especially in the healthcare setting. Early detection of CPE carriage in hospitalized patients with risk factors for CPE carriage is essential to prevent their spread in hospitals as well as to guide empiric antibiotic therapy for CPE carriers with signs of severe infection. However, the prevalence of CPE carriage on admission to hospital is not precisely known, nor are factors associated with CPE carriage.

Hence, the investigators sought to determine the prevalence of CPE carriage and its risk factors in patients admitted to hospital, in order to identify the appropriate indications for CPE screening on admission to hospital. Secondly, the investigators aimed to estimate the annual number of patients with CPE carriage who would not have been identified with the current targeted screening policy as well as to estimate the annual number of secondary cases that could be prevented if a universal screening policy was applied on admission (i.e. for all hospitalized patients, not just those with risk factors).

Therefore, the investigators plan to carry out a systematic screening for rectal carriage of CPE on admission in a sample of patients hospitalized at the Bichat - Claude-Bernard Hospital. Inclusion criteria will include: Age ≥ 18 years, admission to a medical, surgical, obstetrical or intensive care unit at Bichat - Claude-Bernard Hospital in the previous 72 hours, no objection to participating in the study. Rectal swabs will be taken from all included patients for detection of CPE and/or ESBLE. Patients' characteristics, including sociodemographic data, country of birth and residence, clinical ward, current antibiotic treatment and that in the last 3 months, travel abroad and last geographical areas visited, hospitalization in France and abroad, and history of CPE and ESBLE carriage or infection in the previous year, will be collected by questionnaire and from medical records. "

DETAILED DESCRIPTION:
"Introduction The emergence and spread of emerging highly resistant bacteria, including carbapenemase-producing Enterobacteriaceae (CPE), is a public health challenge given their rapid spread and the lack of active antibiotics against these bacteria. The spread of extended-spectrum β-lactamase-producing Enterobacteriaceae (ESBLE) since the early 2000s raises concerns about a potential similar spread of CPE in the coming years, especially in the healthcare setting. Early detection of CPE carriage in hospitalized patients with risk factors for CPE carriage is essential to prevent their spread in hospitals as well as to guide empiric antibiotic therapy for CPE carriers with signs of severe infection. However, the prevalence of CPE carriage on admission to hospital is not precisely known, nor are factors associated with CPE carriage.

Therefore, the investigators plan to carry out a systematic screening for rectal carriage of CPE on admission in a sample of patients hospitalized at the Bichat - Claude-Bernard Hospital.

Primary objective

- To determine the prevalence of CPE carriage in patients admitted to the Bichat - Claude-Bernard Hospital

Secondary objectives

* To determine the prevalence of ESBLE carriage in patients admitted to the Bichat - Claude-Bernard Hospital
* To determine the risk factors for rectal carriage of CPE and ESBLE on admission
* To estimate the annual number of patients with rectal CPE who would not have been identified with the current targeted screening policy
* To estimate the annual number of secondary cases that could be prevented that could be prevented if a universal screening policy was applied on admission (i.e. for all hospitalized patients, not just those with risk factors).
* To characterize the bacterial strains and enzymes identified in CPE carriage on admission.

Materials and methods The study will be performed at a two-site 1000-bed public University Hospital in Paris (France), which provides primary and tertiary care and is located in an area serving a large proportion of foreign-born patients, originating mainly from Africa.

Current criteria for CPE screening on admission to Bichat - Claude-Bernard Hospital include :

* History of hospitalization for more than 24 hours abroad in the last 12 months (since 2010) or
* Travel abroad without hospitalization in the last 12 months, depending on the hospitalization ward and/or the presence of risk factors such as recent return , extended stay or travel in South-East Asia (since 2018)

Rectal swabs will be taken from all included patients by nursing staff or by the patients themselves. Swabs will be discharged on selective media for ESBLE (ChromID ESBLE agar - bioMérieux) and selective media for CPE (chromID® CARBA agar - bioMérieux and chromID® OXA-48TM agar - bioMérieux). An identification by MALDI-TOF mass spectrometry and an antibiogram on Mueller-Hinton agar will be carried out on each suspect colony. A GeneXpert PCR (Cepheid) on suspect colonies will be carried out jointly in the event of a positive culture on selective medium for the detection of CPE. In case of a positive GeneXpert PCR on suspect colonies, a confirmatory GeneXpert PCR will be performed on the native sample.

The following data will be collected from medical records and by questionnaire :

* Socio-demographic characteristics of patients: Age, sex, country of birth, main country of residence, place of residence before hospitalization
* Characteristics of hospital stay: Date of entry into the ward, date of entry into the hospital, origin before admission
* Exposure abroad: Travel/hospitalization abroad in the last 12 months for the patient, travel/hospitalization abroad in the last 12 months for the person(s) living in the same household as the patient
* Exposure to health care facilities: Hospitalization (> 24h) in a health care facility in France in the last 12 months
* Antibiotic exposure: Antibiotic treatment received on the day of the survey or in the previous 3 months
* EBSLE/CPE screening: Known CPE carriage, rectal screening for CPE already taken by the ward healthcare team

The sample size was calculated on a hypothesis of a prevalence of CPE carriage. Assuming a prevalence of 0.5% based on literature data with a 95% confidence interval of [0.1% - 0.9%], 1195 patients should be included. The study will last 6 months with an inclusion period of 6 months; each patient's participation will last 1 day.

The main outcome will be CPE carriage; CPE carriers will be compared with non carriers. Categorical variables will be compared using the Chi-2 test or Fisher's exact test and continuous variables using the Student's t-test or the Mann-Whitney test. Odds ratios (OR) and 95% confidence intervals (CI) will be calculated. All tests will be two-tailed and the significance level will be 5%. The open-source software R for Statistical Computing will be used for the statistical analysis."

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years
* Admission to a medical, surgical, obstetrical or intensive care unit at Bichat - Claude-Bernard Hospital in the previous 72 hours
* No objection to participating in the study

Non-inclusion criteria

* Admission to Bichat - Claude-Bernard Hospital > 72 hours before inclusion
* Readmission to the same ward after discharge
* Hospitalization in a rehabilitation unit or a long-stay unit
* Non affiliation to social security
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to an MCO (Medicine-Surgery-Obstetrics) hospitalization department or intensive care unit at Bichat - Claude-Bernard Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1195 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with CPE carriage | 72 hours

SECONDARY OUTCOMES:
Percentage of patients with ESBLE carriage | The same rectal swab will be used for detection of CPE carriage and ESBLE carriage
  A rectal swab will be taken within 72 hours of admission from a sample of patients admitted to the Bichat - Claude-Bernard Hospital over a 6-month period.
Odds ratios associated with risk factors for CPE and ESBLE carriage on admission to hospital | 6 months after study start
Annual number of patients with rectal CPE carriage among those with no risk factors for CPE carriage | 1 year after study start
Annual number of secondary cases of CPE carriage that could be prevented if a universal admission screening policy was implemented | 1 year after study start
Names and percentages of bacterial species and enzymes identified in CPE screening | 6 months after study start

CONTACTS AND LOCATIONS:
Overall Officials: Solen Kernéis, MD - PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bichat Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No